CLINICAL TRIAL: NCT06708195
Title: Analysis of the Efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) in Patients With Xerostomia
Brief Title: Efficacy of Transcutaneous Electrical Nerve Stimulation in Patients With Xerostomia (ETENX)
Acronym: ETENX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, MD,PhD,DDs, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACTA10/2024/CEI
Record Dates: First submitted 2024-11-20; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Xerostomia; Dry Mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Experimental group Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I :Experimental (Experimental): Patients in this group will receive 15 minutes of extraoral TENS applied to the skin over the bilateral parotid glands. The treatment will consist of 3 sessions per week for 3 weeks.
  Intervention:
  Type: Active TENS Frequency: 3 sessions per week Session duration: 15 minutes Application area: Skin over the bilateral parotid glands
  Interventions: Device: Group experimental
- Control (Sham Comparator): Patients in this group will receive 15 minutes of extraoral TENS applied to the skin over the bilateral parotid glands. However, the device will be inactive ( sham ). This treatment will consist of a single session.
  Intervention:
  Type: Inactive TENS Frequency: 1 session Session duration: 15 minutes Application area: Skin over the bilateral parotid glands
  Interventions: Device: Group experimental

INTERVENTIONS:
Device: Group experimental — Type: Inactive TENS (placebo) Frequency: 1 session Session duration: 15 minutes Application area: Skin over the bilateral parotid glan

SUMMARY:
Saliva is a complex fluid with essential functions in the oral cavity, such as lubricating tissues, protecting against microorganisms, and facilitating processes like chewing, swallowing, and speaking. Xerostomia, defined as the subjective sensation of dry mouth, is commonly associated with reduced salivary flow, which can lead to intraoral and extraoral complications, including dental caries, periodontal disease, infections, and functional difficulties like chewing, speaking, and swallowing.

Current treatments for xerostomia, such as saliva substitutes and lubricants, provide only temporary relief and do not address the underlying cause. Pharmacological agents like pilocarpine have shown effectiveness in stimulating salivary flow; however, their use is limited by adverse side effects such as excessive sweating and gastrointestinal discomfort.

In this context, transcutaneous electrical nerve stimulation (TENS), a physical therapy traditionally used for pain relief, has shown significant potential in the therapeutic stimulation of salivary glands. TENS is a non-invasive approach that works by stimulating the auriculotemporal nerve, which innervates the parotid glands, promoting an increase in salivary flow.

This study highlights the therapeutic value of TENS as an effective and safe solution for patients with xerostomia. The findings indicate that TENS therapy can increase salivary flow, alleviate symptoms of dry mouth, and significantly improve patients' quality of life, all without the risks and adverse effects associated with pharmacological treatments.

DETAILED DESCRIPTION:
Current treatments for xerostomia, such as saliva substitutes and lubricants, provide only temporary relief and do not address the underlying cause. Pharmacological agents like pilocarpine have shown effectiveness in stimulating salivary flow; however, their use is limited by adverse side effects such as excessive sweating and gastrointestinal discomfort.

In this context, transcutaneous electrical nerve stimulation (TENS), a physical therapy traditionally used for pain relief, has shown significant potential in the therapeutic stimulation of salivary glands. TENS is a non-invasive approach that works by stimulating the auriculotemporal nerve, which innervates the parotid glands, promoting an increase in salivary flow.

This study highlights the therapeutic value of TENS as an effective and safe solution for patients with xerostomia. The findings indicate that TENS therapy can increase salivary flow, alleviate symptoms of dry mouth, and significantly improve patients' quality of life,

ELIGIBILITY:
Inclusion Criteria:

Present continuous symptoms of dry mouth for more than three months. Ability to attend the necessary visits to carry out the research.

Exclusion Criteria:

Patient subjected to total or partial resection of major salivary glands. Patient with decompensated systemic disease. Patient who has undergone radiotherapy. Patient with motor impairments or issues preventing them from following the operator's instructions.

Patient with vertigo, persistent headaches, hearing problems, neuralgias, and/or facial paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
The Modified Schirmer tear strip Test measured intensity of salivary flow | Baseline (before the start of each session) and immediately after each session, for a total of 3 sessions over 3 weeks (6 measurements in total: Days 0, 7, and 14).
  Test measured intensity of salivary flow
The Modified Schirmer tear strip Test measured intensity of salivary flow | baseline (day 0 before the start of each session) and immediately after each session, for a total of 3 sessions over 3 weeks (6 measurements in total: Days 0, 7, and 14).
  Test measured intensity of salivary flow
Test Thomson xerostomy | Baseline (day 0 prior to the first session) and at 3 weeks (end of treatment)
  Xerostomia Inventory. the higher the outcome, quality of life decreases
Visual Analogue Scale (VAS) for xerostomia severity | Baseline (day 0 before the start of each session) and immediately after each session, for a total of 3 sessions over 3 weeks (6 measurements in total: Days 0, 7, and 14).
  Visual Analogue Scale (VAS) for xerostomia severity (0 cm: no xerostomía , 10cm : very severe xerostomia ).

SECONDARY OUTCOMES:
OHIP-14 questionnaire | Baseline (day 0) and at 3 weeks (end of treatment)
  Quality of oral life. minimun 0 maximum 56 points. As it gets higher, quality of life decreases

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Khamdi S, Matangkasombut O, Lam-Ubol A. Non-pharmacologic interventions for management of radiation-induced dry mouth: A systematic review. Oral Dis. 2024 Jul;30(5):2876-2893. doi: 10.1111/odi.14804. Epub 2023 Nov 9. PMID 37946598
- [Background] Chandra R, Bhakta P, Beniwal J, Dhanda R, Saxena V, Sinha S. Evaluation of the efficacy of transcutaneous electrical nerve stimulation (TENS) on salivary flow rate in patients with xerostomia - A case control study. J Family Med Prim Care. 2022 Feb;11(2):767-771. doi: 10.4103/jfmpc.jfmpc_922_21. Epub 2022 Feb 16. PMID 35360757
- [Background] Sivaramakrishnan G, Sridharan K. Electrical nerve stimulation for xerostomia: A meta-analysis of randomised controlled trials. J Tradit Complement Med. 2017 Feb 14;7(4):409-413. doi: 10.1016/j.jtcme.2017.01.004. eCollection 2017 Oct. PMID 29034187